CLINICAL TRIAL: NCT05737121
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Multi-Center Single Dose Study to Evaluate the Safety and Effectiveness of VNX001 Compared to Placebo, and the Individual Components of Lidocaine, and Heparin in Subjects With Interstitial Cystitis/Bladder Pain Syndrome Who Have an Episode of Acute Bladder Pain of Moderate to Severe Intensity; The Engage 2024 Study
Brief Title: Safety and Efficacy Study of VNX001 Compared to Its Individual Components (Lidocaine and Heparin) or Placebo in Subjects With IC/BPS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vaneltix Pharma, Inc. (Industry)
Collaborators: Prevail Infoworks (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VNX001-111; Engage 2024
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Interstitial Cystitis; Bladder Pain Syndrome
Keywords: interstitial cystitis (IC); bladder pain syndrome (BPS); alkalinized lidocaine; heparin; intravesical; VNX001
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Heparin; Lidocaine

STUDY DESIGN:
Intervention Model Description: IC/BPS patients will be randomly assigned to receive a single dose of one of the following treatments in a ratio of 3:1:3:1:
  * VNX001 (n=45): alkalinized buffered lidocaine HCl (200 mg) and heparin sodium (50,000 USPU), administered as an intravesical instillation
  * Placebo (n=15): alkalinized buffer, administered as an intravesical instillation
  * Lidocaine (n=45): alkalinized buffered lidocaine HCl (200 mg), administered as an intravesical instillation
  * Heparin (n=15): alkalinized buffered heparin sodium (50,000 USPU), administered as an intravesical instillation
  * At 24-48-hours post-dose, all subjects will be given the option of requesting a single open-label dose of VNX001.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- VNX001 (Experimental): VNX001 (lidocaine HCl [200 mg] and heparin sodium [50,000 USPU] in alkalinized buffer), administered as a single dose via intravesical instillation; n=45 (anticipated)
  Interventions: Drug: VNX001
- Placebo (Placebo Comparator): Alkalinized buffer, administered as a single dose via intravesical instillation; n=15 (anticipated)
  Interventions: Drug: Placebo
- Lidocaine (Experimental): Lidocaine HCl (200 mg) in alkalinized buffer, administered as a single dose via intravesical instillation; n=45 (anticipated)
  Interventions: Drug: Lidocaine
- Heparin (Experimental): Heparin sodium (50,000 USPU) in alkalinized buffer, administered as a single dose via intravesical instillation; n=15 (anticipated)
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: VNX001 — VNX001 (alkalinized lidocaine HCl and heparin sodium)
  Other Names: Alkalinized lidocaine HCl and heparin sodium
  Arms: VNX001
Drug: Placebo — Inactive placebo for VNX001
  Other Names: Placebo (for VNX001)
  Arms: Placebo
Drug: Lidocaine — Alkalinized lidocaine hydrochloride
  Other Names: Alkalinized lidocaine HCl
  Arms: Lidocaine
Drug: Heparin — Alkalinized heparin sodium
  Other Names: Alkalinized heparin sodium
  Arms: Heparin

SUMMARY:
This is a Phase 2, prospective, randomized, double-blind, placebo-controlled, multi-center, single-dose, pharmacodynamic study designed to evaluate the efficacy and safety of the combination product (VNX001) versus placebo and its individual components (heparin sodium and lidocaine hydrochloride (HCl)) for the reduction of bladder pain in patients with interstitial cystitis (IC) / bladder pain syndrome (BPS), Who Have an Episode of Acute Bladder Pain of Moderate to Severe Intensity.

DETAILED DESCRIPTION:
This is a Phase 2, prospective, randomized, double-blind, placebo-controlled, multi-center, single-dose, pharmacodynamic study designed to evaluate the efficacy and safety of the combination product (VNX001) versus placebo and its individual components (heparin sodium and lidocaine hydrochloride) for the reduction of bladder pain in patients with IC/BPS, Who Have an Episode of Acute Bladder Pain of Moderate to Severe Intensity. The study will enroll a target of 120 subjects, with a maximum of 180 subjects, across approximately 12 sites in the United States. Each study subject will receive a single dose of VNX001, placebo (alkalinized phosphate buffer), alkalinized lidocaine, or alkalinized heparin by random assignment. The randomization ratio will be 3:1:3:1, respectively. At 24-48-hours post-dose, all subjects will be given the option of requesting a single dose of VNX001.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to give a signed informed consent and to follow study instructions
* Be male or female, ≥ 18 years of age
* Have a history of IC/BPS for at least 9 months prior to the study
* Have a score of ≥ 16 and ≤ 30 on the Pelvic Pain and Urgency/Frequency (PUF) questionnaire, completed at screening
* Have an episode of acute bladder pain of moderate to severe intensity with a minimum score of 5 on the 11-point bladder pain NRS at time of screening and 15 minutes post void immediately prior to study drug administration.
* Have previously received a therapeutic intravesicular anesthetic treatment according to medication history

Exclusion Criteria:

* For females, have a positive pregnancy test at screening or be pregnant or lactating
* Males who are sexually active with females and are not willing to commit to an acceptable method of birth control for the duration of the
* Postmenopausal women who, if taking hormone replacement therapy, have not been stabilized on a regimen of hormone replacement therapy within 3 months of screening
* Have a known hypersensitivity to heparin or lidocaine
* Have used any local anesthetic by any route within 48-hours prior to study drug administration, or used a lidocaine patch or lidocaine containing topical compounds within 14 days prior to study drug administration
* Have used a tricyclic antidepressant, or a gamma-aminobutyric acid (GABA) analogue (gabapentin or pregabalin), unless taking a stable dose of the medication for ≥ 3 weeks. The stable dose of gabapentin may not exceed 1,200 mg per day, and the stable dose of pregabalin may not exceed 150 mg per day
* Have used any pain medication within 6 hours prior to study drug administration
* Have used narcotics or medical marijuana ≤ 3 weeks prior to study entry
* Have used prohibited drugs as determined by self-report, positive urine drug screen, or in the opinion of the investigator be under the influence of drugs affecting mentation precluding their ability to follow the study protocol or bias study results
* Have a known abnormal laboratory test value that, in the investigator's judgement, is clinically significant.
* Have a neurogenic bladder or other disorder that, in the opinion of the investigator, may cause neurogenic bladder (including Parkinson's disease, multiple sclerosis, epilepsy, myasthenia gravis, movement disorders, spinal cord damage)
* Have pain or a pain disorder that, in the opinion of the investigator, would make it difficult to discriminate pelvic pain of bladder origin from the other pain
* Have any of the following central nervous system (CNS) conditions that in the opinion of the investigator would impact the subject's study participation due to their ability to follow the study protocol or bias study results, severe diagnosed: major depressive disorder, bipolar disorder, schizophrenia, general anxiety disorder, attention deficit disorder, obsessive compulsive disorder, or other major central nervous system disorder
* Have history of arrhythmias, conduction disturbances, or cardiac disease, or any coexisting medical condition that, in the opinion of the investigator, may be significant or interfere with study procedures or interpretation of study results
* Had anesthetic bladder instillation therapy within 14 days prior to study entry
* Had an in-office cystoscopy within 7 days of study drug administration
* Had dilatation (hydrodistension) of bladder within 3 months of study entry
* Evidence or suspected presence of cancer detected during cystoscopy 7 days prior to or at time of initial screening
* Has received any investigational drug or device within 30 days prior to screening
* Is currently enrolled in another investigational drug or device study
* Is unwilling or unable to abide by the requirements of the study
* Have an actively bleeding lesion or area in the bladder as detected by dipstick urinalysis and investigator assessment, immediately prior to randomization
* Have a history of coagulopathy or taking anticoagulants.
* Are taking any of the following medications, which are inducers of CYP1A2 and/or CYP3A4: Phenytoin, Carbamazepine, St. John's Wort, Phenobarbital, Rifampin
* Have had any of the following:

  * Bacterial cystitis within 30 days as demonstrated by a positive urine culture (≥ 105 bacteria per mL)
  * History of pelvic irradiation or radiation cystitis
  * History or presence of uterine, cervical, pelvic, rectal, ovarian, or vaginal cancer
  * History of benign or malignant bladder tumors
  * Current chemotherapy
  * History or presence of tuberculous cystitis
  * History or presence of chemical cystitis, including that due to cyclophosphamide
  * History or presence of urinary schistosomiasis
  * Bladder or ureteral calculi
  * Clinically significant infectious vaginitis
  * Currently uncontrolled genital herpes
  * History or presence of urethral diverticulum
  * Presence of bladder fistulae
  * History of ketamine use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Sum of bladder pain intensity differences from baseline to 12 hours post-dose (SPID-12) | 12 hours
  A measure of the sum of bladder pain intensity differences from baseline to 12 hours post-dose (SPID-12), as determined using an 11-point numerical rating scale (NRS) for bladder pain. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.

SECONDARY OUTCOMES:
Sum of bladder pain intensity differences from baseline to 6, 10, and 24 hours post-dose (SPID-6, SPID-10, and SPID-24, respectively) | 6, 10, or 24 hours
  A measure of the sum of bladder pain intensity differences from baseline to 6, 10, and 24 hours post-dose (SPID-6, SPID-10, and SPID-24, respectively), as determined using an 11-point numerical rating scale (NRS) for bladder pain. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Change in bladder pain from baseline to 1, 4, 8, 12, and 24 hours post-dose | 1, 4, 8, 12, and 24 hours
  Average absolute change and average percentage change in bladder pain from baseline to 1, 4, 8, 12, and 24 hours post-dose, as determined using an 11-point numerical rating scale (NRS) for bladder pain. The 11-point NRS for bladder pain is a scale from 0 to 10, with 0 indicating no bladder pain and 10 indicating the worst imaginable bladder pain.
Change in Question 3 of the Patient Overall Rating of Improvement of Symptoms (PORIS) questionnaire | 1, 10, and 24 hours
  Percentage of subjects achieving ≥ 50% improvement in Question 3 of the PORIS questionnaire at 1, 10, and 24 hours post-dose. The PORIS questionnaire is an assessment of the subject's condition after treatment compared to before treatment. In particular, Question 3 of the PORIS questionnaire asks subjects to select the category that best describes the overall change in their condition compared to before receiving study medication; the choices are: worse, no better (0% improvement), slightly improved (25% improvement), moderately improved (50% improvement), greatly improved (75% improvement), or symptoms gone (100% improvement).
Use of optional open-label intravesical administration of VNX001 | 48 hours
  Number of patients requesting the optional open-label intravesical administration of VNX001 at 24-48 hours after randomized study drug administration
Adverse events (AEs) | 72 hours
  Incidence of treatment-emergent adverse events (TEAEs), drug-related adverse events (AEs), and discontinuations due to AEs

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - IC Study LLC, Escondido, California
  - University of California Los Angeles Center for Women's Pelvic Health, Los Angeles, California
  - The Clark Center for Urogynecology, Newport Beach, California
  - The Continence Center Medical Group, Inc dba Southern California Continence Center, Newport Beach, California
  - University of California San Diego Medical Center, San Diego, California
  - Prestige Medical Group, Tustin, California
  - United Research Institute, Hialeah, Florida
  - Florida Urology Partners, Tampa, Florida
  - Georgia Urology, Cartersville, Georgia
  - Southern Clinical Research Associates LLC, Metairie, Louisiana
  - Bay State Clinical Trials, Watertown, Massachusetts
  - Sheldon Freedman MD LTD, Las Vegas, Nevada
  - Northwell Health, Lake Success, New York
  - The Wake Forest Institute of Regenerative Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ENGAGE2024 Study Website — https://engage-24.com/